CLINICAL TRIAL: NCT02460666
Title: Brain Connectivity and Response to Tai Chi in Geriatric Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01AT008383-01A1 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-06-02 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
Keywords: depressed; older adults; Major Depressive Disorder; Tai-Chi; geriatric
MeSH Terms: conditions — Depressive Disorder, Major; Consciousness Disorders | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai-Chi Chih Classes (Experimental): Participants will engage in 12 weekly 60 minute Tai-Chi-Chih classes.
  Interventions: Behavioral: Tai-Chi-Chih (TCC)
- Health Education and Wellness Classes (Active Comparator): Participants will engage in 12 weekly 60 minute Health Education and Wellness classes.
  Interventions: Behavioral: Health Education and Wellness Classes (HEW)

INTERVENTIONS:
Behavioral: Tai-Chi-Chih (TCC)
  Other Names: Tai Chi
  Arms: Tai-Chi Chih Classes
Behavioral: Health Education and Wellness Classes (HEW)
  Arms: Health Education and Wellness Classes

SUMMARY:
The purpose of this study is to evaluate the effects after up to 1 year of supervised weekly Tai-Chi-Chi versus Health Education and Wellness classes on reduction of depressive symptoms and improvement in resilience, health functioning, quality of life, cognition, sleep, fMRI neural correlates of working memory, and brain structure.

DETAILED DESCRIPTION:
The proposed randomized trial aims to investigate neural mechanisms of brain connectivity when comparing response to TCC to health and wellness education classes using fMRI biomarkers of emotional regulation and cognition. Control group will include health wellness education programs (HEW) that will help to control for the non-specific social support factors. Primary outcomes include measures of depressive symptom severity. Secondary outcomes include cognition, resilience, health functioning, quality of life. Maintenance of response and relapse of major depression will be determined during 6 month (and 12 month follow-up if MRI eligible). Functional magnetic resonance imaging (fMRI) correlates of emotional processing and connectivity in related functional networks. Neural correlates of working memory, and brain structure will be examined in ½ of the sample. The researchers will investigate whether variations in emotional regulation will moderate or predict emotional and functional improvement linked to TCC.

The investigators will recruit 220 older adults with depressive symptoms who have been on a stable form of treatment for at least 4 months, who will be randomly assigned to 12 weeks of: 1.Ta-Chi-Chih (TCC) class; or 2. Health/Wellness Education Program (HEW); all for 120 minutes per week. All subjects will receive comprehensive evaluations of mood, mental and physical health, and cognition at baseline, 12 weeks, and 6 months. Changes over time in measures of depressive symptoms, resilience, quality of life, and cognition will be assessed in random regression models. The investigators anticipate that greater clinical improvement in mood and cognition will in the TCC group compared to the HEW. The investigators also expect clinical improvement to correlate with the change in the activation in the right ventrolateral prefrontal cortex (VLPFC) and amygdala in an affect labeling task, and working memory-related activation of dorsolateral prefrontal cortex (DLPFC), and change in functional connectivity in brain network activity. This is the first randomized trial of response to TCC that integrates the use of fMRI biomarkers of response to guide the development of treatment and preventive approaches in geriatric depression.

ELIGIBILITY:
Inclusion Criteria:

* A 24-item Hamilton Rating Scale for Depression (HAMD) score greater than 14 consistent with moderate-severe depression.
* Mini-Mental State Exam (MMSE) score greater than 24.
* Sufficient English proficiency and 8th grade or higher reading level as determined by the word reading subtest of the Wide Range Achievement Test-IV.
* Capacity to provide informed consent.
* A stable form of treatment for at least 4 months.

Exclusion Criteria:

* Any current or past psychiatric disorders, or recent unstable medical or neurological disorders
* Any disabilities preventing their participation in Tai-Chi Chih exercise (e.g. severe visual or hearing impairment)
* Insufficient English proficiency
* Diagnosis of dementia
* Mini Mental Health Examination score of 24 and below
* Effective antidepressant, psychotropic medications, or effective therapy
* Participation in a psychotherapy that involves cognitive training
* Do not meet criteria for moderate-severe depression with a 24-item Hamilton Rating Scale for Depression (HAMD) score less than 14

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01; Primary Completion 2020-11-18 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin MR, Olmstead R, Carrillo C, Sadeghi N, Breen EC, Witarama T, Yokomizo M, Lavretsky H, Carroll JE, Motivala SJ, Bootzin R, Nicassio P. Cognitive behavioral therapy vs. Tai Chi for late life insomnia and inflammatory risk: a randomized controlled comparative efficacy trial. Sleep. 2014 Sep 1;37(9):1543-52. doi: 10.5665/sleep.4008. PMID 25142571
- [Background] Siddarth D, Siddarth P, Lavretsky H. An observational study of the health benefits of yoga or tai chi compared with aerobic exercise in community-dwelling middle-aged and older adults. Am J Geriatr Psychiatry. 2014 Mar;22(3):272-3. doi: 10.1016/j.jagp.2013.01.065. Epub 2013 May 2. No abstract available. PMID 23642461
- [Background] Lavretsky H, Alstein LL, Olmstead RE, Ercoli LM, Riparetti-Brown M, Cyr NS, Irwin MR. Complementary use of tai chi chih augments escitalopram treatment of geriatric depression: a randomized controlled trial. Am J Geriatr Psychiatry. 2011 Oct;19(10):839-50. doi: 10.1097/JGP.0b013e31820ee9ef. PMID 21358389
- [Background] Schneider B, Ercoli L, Siddarth P, Lavretsky H. Vascular burden and cognitive functioning in depressed older adults. Am J Geriatr Psychiatry. 2012 Aug;20(8):673-81. doi: 10.1097/JGP.0b013e31822ccd64. PMID 21857219
- [Background] Abbott R, Lavretsky H. Tai Chi and Qigong for the treatment and prevention of mental disorders. Psychiatr Clin North Am. 2013 Mar;36(1):109-19. doi: 10.1016/j.psc.2013.01.011. PMID 23538081
- [Derived] Lavretsky H, Milillo MM, Kilpatrick L, Grzenda A, Wu P, Nguyen SA, Ercoli LM, Siddarth P. A Randomized Controlled Trial of Tai Chi Chih or Health Education for Geriatric Depression. Am J Geriatr Psychiatry. 2022 Mar;30(3):392-403. doi: 10.1016/j.jagp.2021.07.008. Epub 2021 Jul 30. PMID 34404606

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 220 participants were enrolled after providing consent and completing the screen visit. 178 participants completed baseline procedures and were randomized to either group.
Groups:
- Tai-Chi Chih Classes: Participants will engage in 12 weekly 60 minute Tai-Chi-Chih classes.
  Tai-Chi-Chih (TCC)
- Health Education and Wellness Classes: Participants will engage in 12 weekly 60 minute Health Education and Wellness classes.
  Health Education and Wellness Classes (HEW)
Period: Overall Study
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Started | 89 | 89
Completed | 62 | 63
Not Completed | 27 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (6.9) | 69.4 (6.2) | 69.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 27 | 22 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 83 | 85 | 168
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 76 | 77 | 153
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 89 | 89 | 178
Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Clinician administered scale measures severity of depressive symptoms. This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
  units on a scale | 19.0 (4.0) | 19.3 (3.9) | 19.15 (3.91)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HDRS) Scores
Description: Clinician administered scale measures severity of depressive symptoms. This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
Time Frame: Measured at baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Number analyzed (Participants) | 62 | 63
units on a scale | -9.27 (5.29) | -9.40 (5.35)
Statistical Analysis 1: Comparison: Tai-Chi Chih Classes vs Health Education and Wellness Classes; Test type: Superiority; p = 0.3, Mixed Models Analysis

2. Secondary Outcome: Change in Delayed Recall Cognitive Domain Scores
Description: Neuropsychological battery of tests which included the following domains:
  Delayed Recall (CVLT-II [Long-Delay Free Recall], Rey-Osterrieth Complex Figure Test [30-minute Delayed Recall])
  Raw scores were transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across both arms) is zero for each test score. These z-scores were then averaged within each neuropsychological domain to produce composite scores. Higher scores are indicative of better performance.
Time Frame: Measured at baseline and 3 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Number analyzed (Participants) | 62 | 63
z-score | -0.15 (0.57) | -0.002 (0.61)
Statistical Analysis 1: Comparison: Tai-Chi Chih Classes vs Health Education and Wellness Classes; Test type: Superiority; p = 0.2, Mixed Models Analysis

3. Secondary Outcome: Change in Attention/Executive Function Cognitive Domain Scores
Description: Neuropsychological battery of tests which included the following domains:
  Attention/Executive Function (Trail Making Test A and B, Stroop Interference [Golden version])
  Raw scores were transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across both arms) is zero for each test score. These z-scores were then averaged within each neuropsychological domain to produce composite scores. Higher scores are indicative of better performance.
Time Frame: Measured at baseline and 3 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Number analyzed (Participants) | 62 | 63
z-score | -0.04 (0.61) | 0.03 (0.53)
Statistical Analysis 1: Comparison: Tai-Chi Chih Classes vs Health Education and Wellness Classes; Test type: Superiority; p = 0.5, Mixed Models Analysis

4. Secondary Outcome: Change in Language Cognitive Domain Scores
Description: Neuropsychological battery of tests which included the following domains:
  Language (Controlled Oral Word Association test [FAS], Animal Fluency, and Boston Naming Test)
  Raw scores were transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across both arms) is zero for each test score. These z-scores were then averaged within each neuropsychological domain to produce composite scores. Higher scores are indicative of better performance.
Time Frame: Measured at baseline and 3 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Number analyzed (Participants) | 62 | 63
z-score | 0.03 (0.40) | -0.12 (0.46)
Statistical Analysis 1: Comparison: Tai-Chi Chih Classes vs Health Education and Wellness Classes; Test type: Superiority; p = 0.09, Mixed Models Analysis

5. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: The UKU (Udvalg for Kliniske Undersogelser) Side Effect Rating Scale organizes symptoms into 4 categories (i.e., Psychic, Neurologic, Autonomic, Other) containing 8-19 symptoms each. Each symptom receives a score for degree and causal relationship. Degree is scored between 0-3 with higher scores being more severe. Causal relationship is scored as improbable, possible, or probable.
Time Frame: Measured at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
Number analyzed (Participants) | 89 | 89
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of 6 months, from the time the participants began the intervention until the Week 24 follow-up.
Description: Adverse events were obtained via the UKU Side Effect Rating Scale, where items were scored on a 0-3 scale for degree (0 = none, 1 = mild, 2 = moderate, 3 = severe) and on a scale of 1-3 of probability if an adverse event was present (1 = impossibly related, 2 = possibly related, 3 = probably related).
Arm/Group | Tai-Chi Chih Classes | Health Education and Wellness Classes
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 4/89 | 3/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai-Chi Chih Classes (N=89) | Health Education and Wellness Classes (N=89)
Asthenia/Lassitude/Increased Fatigability (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Failing memory (Psychiatric disorders) | 0 (0) | 1 (1)
Tension/Inner Unrest (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
After March 18th, 2020, all assessments were completed remotely due to COVID-19 until restrictions were lifted for eligible participants to come in-person.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT02460666/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02460666/ICF_000.pdf